CLINICAL TRIAL: NCT00188110
Title: Evaluation of the Water-Enema Computed Tomography for the Diagnosis of Colon Tumor
Brief Title: Performance of the Water-Enema Computed Tomography (WE-CT)
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: University Hospital, Angers (Other Government)
Collaborators: Ministry of Health, France (Other Government)
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: PHRC-02-01; 2002/23 (CCPPRB)
Record Dates: First submitted 2005-09-12; First posted 2005-09-16 (Estimated); Last update posted 2007-01-09 (Estimated); Status verified 2005-09

CONDITIONS: Colon Cancer
Keywords: Water-Enema Computed Tomography; colon tumor; coloscopy; suspicion of colon tumor; coloscopy or surgery
MeSH Terms: conditions — Colonic Neoplasms

INTERVENTIONS:
Procedure: Water-Enema Computed Tomography

SUMMARY:
The WE-CT is an innovative and easy practice imaging technique of colon tumors; it is based on the colon distension by a high volume of warm water and a multidetector CT acquisition after IV (intravenous) contrast, allowing image analysis including the wall thickness and enhancement, the pericolic adjacent spaces and the entire abdomen.

The goal of the study is the evaluation of its performances for the diagnosis of colon tumors.

ELIGIBILITY:
Inclusion Criteria:

* Written informed consent
* WE-TC indication for colon tumor suspicion
* Age > 18 years

Exclusion Criteria:

* Pregnancy
* Patients under 65 years old and for whom the only WE-TC indication is familial antecedents of colon tumor, without clinical or para-clinical personal signs for this pathology
* Infected sigmoid diverticulosis
* Occlusive syndrome
* Anesthesia contraindications
* Anal incontinence
* Renal insufficiency (creatinine > 150 micromol/L)
* Iode allergy
* Visceralgine contraindications
* Scania contraindications

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 200
Dates: Start 2003-03

PRIMARY OUTCOMES:
To evaluate the performances of the WE-CT in patients suspected of having a colon tumor

SECONDARY OUTCOMES:
To show the CT findings in case of colon tumor and its pitfalls
To demonstrate the advantages of the WE-CT compared to the CT and magnetic resonance (MR) colonography for the diagnosis and local staging of colon tumors

CONTACTS AND LOCATIONS:
Overall Officials: Christophe Aube, MD, Principal Investigator — UH of Angers
Locations (5):
- France (5):
  - UH of Angers, Angers
  - UH of Besancon, Besançon
  - UH of Lyon, Lyon
  - UH of Montpellier, Montpellier
  - UH of Rennes, Rennes